CLINICAL TRIAL: NCT01901614
Title: RANDOMIZED CLINICAL TRIAL OF OCT-GUIDED LASER-ASSISTED LAMELLAR ANTERIOR KERATOPLASTY IN ADULTS FOR KERATOCONUS
Brief Title: OCT-guided LALAK for KCN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modifying procedure
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Winston Chamberlain, MD, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU IRB00009280- PTK; R01EY018184 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Corneal Opacity; Keratoconus
Keywords: Keratoconus; Corneal Opacity; Keratoplasty
MeSH Terms: conditions — Corneal Opacity; Keratoconus | interventions — Anesthesia, General; Tomography, Optical Coherence; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LALAK (Experimental): laser-assisted lamellar anterior keratoplasty. Optical Coherence Tomography, femtosecond laser, topical anesthesia, and Retrobulbar Block or General Anesthesia will be used.
  Interventions: Procedure: LALAK; Device: optical coherence tomography (OCT); Drug: Topical Anesthesia; Device: femtosecond laser
- IEK (Active Comparator): Intralase-enabled keratoplasty. Femtosecond laser and Retrobulbar Block or General Anesthesia will be used.
  Interventions: Procedure: IEK; Drug: Retrobulbar Block or General Anesthesia; Device: femtosecond laser

INTERVENTIONS:
Procedure: LALAK — 1. A "dovetail" shaped cut will be made on the graft using a femtosecond laser at the eye bank. The cut depth will be proportional to the central stromal thickness of the graft. This graft will be separated from stromal bed by eye bank personnel for examination of the cut surface. High-quality graft will be replaced in preservation medium and shipped to the surgeon prior to surgery.
  2. The host cornea will receive femtosecond laser cut consisting of a shallow lamellar cut with angled side cut to match the dovetail graft in a tongue-in-groove fashion. The femtosecond laser treatments will be performed under topical anesthesia in the laser suite. The femtosecond laser is an FDA-approved device for use in this indication (corneal transplantation including lamellar keratoplasty). A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Arms: LALAK
Procedure: IEK — 1. A full thickness graft will be prepared at the eye bank with zigzag side cuts prepared with a femtosecond laser. The graft is separated from the rim, replaced in the preservation medium, and shipped to the surgeon prior to the surgery.
  2. In the laser suite, the host cornea will be cut with the femtosecond laser with zigzag side cuts leaving a 70-100 micron bridge. A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Arms: IEK
Drug: Retrobulbar Block or General Anesthesia
  Arms: IEK
Device: optical coherence tomography (OCT) — OCT will be used to guide the depth of the graft and donor dissections.
  Arms: LALAK
Drug: Topical Anesthesia
  Arms: LALAK
Device: femtosecond laser — The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA). The iFS is FDA-approved for corneal surgery including full thickness and lamellar keratoplasty. Eye banks use earlier versions of the Intralase system which are also FDA approved for this indication.

SUMMARY:
The purpose of this study is to determine if a new procedure, called laser-assisted lamellar anterior keratoplasty (LALAK), can achieve the same level of vision with a lower risk of potential complications after surgery compared to another corneal transplant procedure. The current procedure is called Intralase-enabled keratoplasty (IEK) and replaces the entire cornea.

The LALAK procedure involves transplanting only the top layers of the cornea instead of the entire cornea. Only one eye will have this experimental procedure performed. If both eyes need to have surgery your doctor will help you decide on the best non-study option for your other eye.

DETAILED DESCRIPTION:
Corneal transplantation (keratoplasty) is the most common organ transplant, with 42,606 procedures in the U.S. in 2009. Many surgeons are moving away from full thickness corneal transplantation, also called penetrating keratoplasty (PK), because of risks involving rejection, irregular astigmatism and wound dehiscence. They are moving towards partial thickness (lamellar) transplantations of either the anterior or posterior (endothelial) layers, which can reduce these risks.

The femtosecond laser has been used to create excellent tongue-in-groove junctions between the graft and host in full thickness PK.1 This technique, called IEK (Intralase-enabled keratoplasty), has now become a standard surgical procedure. The tongue-in-groove junction achieved at the circumferential edge of the graft and host leads to a continuous smooth anterior surface and strong wound healing.

The new technique is called dovetail LALAK. In this technique, the femtosecond laser is used to create a 31% anterior lamellar graft with dove tailed side cuts. It is also used to create a shallow anterior lamellar dissection and beveled side cuts on the recipient cornea to match with the dovetail graft.

In the new technique, the depth of the graft and donor dissections will be guided by OCT measurements. The proposed trial will test if the new technique can reproducibly achieve good visual outcomes without the risk of rejection. The outcome of the LALAK procedure will be compared to that of IEK.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with keratoconus that cannot be adequately or safely corrected with spectacles, contact lens or excimer laser surface ablation. The cornea must have healthy endothelium (endothelial cell density > 1,500/mm2).

Exclusion Criteria:

1. Preoperative corneal thickness less than 400 microns.
2. Corneal edema
3. Central guttata
4. Inability to give informed consent.
5. Inability to maintain stable fixation for OCT imaging.
6. Inability to commit to required visits to complete the study.
7. Eyes with concurrent cataract, retinal diseases, glaucoma, or other eye conditions that may limit the visual outcome after surgery.
8. Patients with severe collagen vascular diseases or ocular surface disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winston Chamberlain, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: Related Info — http://www.coollab.net

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser-assisted Lamellar Anterior Keratoplasty: Laser-assisted lamellar anterior keratoplasty
  LALAK: a. A "dovetail" shaped cut will be made on the graft using a femtosecond laser at the eye bank. The cut depth will be proportional to the central stromal thickness of the graft. This graft will be separated from stromal bed by eye bank personnel for examination of the cut surface.
  b. The host cornea will receive femtosecond laser cut consisting of a shallow lamellar cut with angled side cut to match the dovetail graft in a tongue-in-groove fashion. The FDA-approved femtosecond laser treatments will be performed under topical anesthesia in the laser suite.
  optical coherence tomography (OCT): OCT will be used to guide the depth of the graft and donor dissections.
  Topical Anesthesia
  femtosecond laser: The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA).
- Intralase-enabled Keratoplasty: Intralase-enabled keratoplasty.
  IEK: a. A full thickness graft will be prepared at the eye bank with zigzag side cuts prepared with a femtosecond laser. The graft is separated from the rim, replaced in the preservation medium, and shipped to the surgeon prior to the surgery.
  b. In the laser suite, the host cornea will be cut with the femtosecond laser with zigzag side cuts leaving a 70-100 micron bridge. A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Retrobulbar Block or General Anesthesia
  femtosecond laser: The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA). The iFS is FDA-approved for corneal surgery including full thickness and lamellar keratoplasty. Eye banks use earlier versions of the Intralase system which are also FDA approved for this indication.
Period: Overall Study
Arm/Group | Laser-assisted Lamellar Anterior Keratoplasty | Intralase-enabled Keratoplasty
Started | 3 | 2
Completed | 1 | 1
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Screen Fail | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Laser-assisted Lamellar Anterior Keratoplasty: LALAK: a. A "dovetail" shaped cut will be made on the graft using a femtosecond laser at the eye bank. The cut depth will be proportional to the central stromal thickness of the graft. This graft will be separated from stromal bed by eye bank personnel for examination of the cut surface.
  b. The host cornea will receive femtosecond laser cut consisting of a shallow lamellar cut with angled side cut to match the dovetail graft in a tongue-in-groove fashion. The FDA-approved femtosecond laser treatments will be performed under topical anesthesia in the laser suite.
  optical coherence tomography (OCT): OCT will be used to guide the depth of the graft and donor dissections.
  Topical Anesthesia
  femtosecond laser: The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA). The iFS is FDA-approved for corneal surgery including full thickness and lamellar keratoplasty.
- Intralase-enabled Keratoplasty: IEK: a. A full thickness graft will be prepared at the eye bank with zigzag side cuts prepared with a femtosecond laser. The graft is separated from the rim, replaced in the preservation medium, and shipped to the surgeon prior to the surgery.
  b. In the laser suite, the host cornea will be cut with the femtosecond laser with zigzag side cuts leaving a 70-100 micron bridge. A protective eye shield is placed over the eye. The graft will be sutured into the host bed.
  Retrobulbar Block or General Anesthesia
  femtosecond laser: The femtosecond laser system to be used in this study for host cornea preparation will be the Intralase FS system (iFS, AMO, Inc., Santa Ana, CA). The iFS is FDA-approved for corneal surgery including full thickness and lamellar keratoplasty. Eye banks use earlier versions of the Intralase system which are also FDA approved for this indication.
- Total: Total of all reporting groups
Arm/Group | Laser-assisted Lamellar Anterior Keratoplasty | Intralase-enabled Keratoplasty | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Does LALAK Achieve the Same Level of Post-operative BSCVA as IEK.
Description: The primary goal of the trial is to determine if LALAK can achieve the same level of postoperative Best Spectacle Corrected Visual Acuity (BSCVA) guided by OCT as IEK. The BSCVA will be measured using a clinic Snellen chart and recorded in the typical Snellen fraction (20/xx) in feet. This will be converted to logMAR form for statistical analysis.
Time Frame: 24 months
Population: For the LALAK group, there were 3 subjects enrolled, but one was a screen fail so no data was obtained for that subject.
Measure: Mean (95% Confidence Interval); unit: logMAR unit
Arm/Group | Laser-assisted Lamellar Anterior Keratoplasty | Intralase-enabled Keratoplasty
Number analyzed (Participants) | 2 | 2
logMAR unit | 0.7 [0.7 to 0.7] | 0.05 [-0.5853 to 0.6853]

ADVERSE EVENTS:
Time Frame: Data was collected up to 24-months from the date of surgery.
Description: See data tables for adverse event information.
Arm/Group | Laser-assisted Lamellar Anterior Keratoplasty | Intralase-enabled Keratoplasty
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser-assisted Lamellar Anterior Keratoplasty (N=2) | Intralase-enabled Keratoplasty (N=2)
Revert to keratoconus pattern (Eye disorders) | 1 (1) | 0 (0)
Corneal epithelial defect with interface haze (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT01901614/Prot_SAP_000.pdf